CLINICAL TRIAL: NCT04090489
Title: Post Treatment Evaluation of Terapeutic Response Biomarkers. Cardiological Studies in Children Treated for Chagas Disease
Brief Title: Congenital Chagas Disease: Long Term Follow up of Treated Children. Preliminary Report or Cardiological Evaluation in Chagas Disease Treated Children
Status: Completed | Type: Observational
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Dr Jaime Altcheh, Principal Investigator, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: Holter Chagas Children
Record Dates: First submitted 2019-09-10; First posted 2019-09-16 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chagas Disease; Chagas Cardiomyopathy
MeSH Terms: conditions — Chagas Disease; Chagas Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chagas disease (CD) could be acquired by contact with the vector, transplacentally and by blood transfusion. The duration and clinical presentation of the initial acute phase of the infection may be variable, but the majority of patients are asymptomatic. The acute phase usually lasts a few months and, if untreated, the acute phase goes on to develop a chronic infection. The chronic phase usually continues for the subject's lifetime, and 30% to 40% of patients will progress to the chronic phase with a cardiac, digestive, neurological, or mixed form at 15 to 30 years after the initial infection. Progressive heart failure and sudden death due to ventricular arrhythmias are the main causes of death in patients with chronic Chagas heart disease.

Objective: To evaluate cardiac involvement in children after pharmacological treatment for Chagas disease.

Methods: Open exploratory study, blind for cardiological evaluation. Population: children treated for Chagas disease with at least 6 years after-treatment parasitological (T.cruzi qPCR), serological (IHA, EIA) and cardiological follow-up. Non-infected subjects were included as a control group for final cardiological evaluation.

Treatment: benznidazole or nifurtimox, standard dose, for 60 days. Blood samples were collected at diagnosis, end-of-treatment and every 6-12 months thereafter.

Electrocardiogram (ECG) was performed at diagnosis and every year after treatment.

In this cohort, 24 hours ECG (Holter) and Speckle-tracking strain echocardiography study were performed at the end of follow-up for this study.

ELIGIBILITY:
Inclusion Criteria:

* Chagas diseases children treated with benznidazole / or nifurtimox
* Patients with at least 6 years of after-treatment follow-up.
* Diagnosis of Chagas disease: in infants younger than 8 months by direct observation of T.cruzi using parasitological concentration method (microhematocrit test); in infants older than 9 months 2 reactive serological test (ELISA, Indirect Hemagglutination ).

Exclusion Criteria:

* Patients with chronic diseases (renal, hepatic, neurological) that at the discretion of the researcher could affect the interpretation of the results.
* Subjects with congenital heart disease.

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A cohort of CD treated children with at least 6 years post-treatment parasitological (T. cruzi qPCR), serological and cardiological follow-up. Treatment: benznidazole (Bz) or nifurtimox (Nftx), standard dose, for 60 days.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of CD treatment in preventing the development of cardiac alterations in treated children. | 10 years
  To compare number of patients with pathological cardiac findings, measured by Holter and ECG, in two different groups: patients with treated Chagas disease (either with Nifurtimox or Benznidazole) and healthy (without Chagas disease) patients of the same population (control group).

SECONDARY OUTCOMES:
Post treatment evaluation of treatment response biomarkers | 5 years
  To compare serology titles in patients treated for Chagas disease (either with Nifurtimox or Benznidazole) with PCR titles in the same group of patients and evaluate if PCR can be an early marker of therapeutic response compared to serology.

CONTACTS AND LOCATIONS:
Locations (1):
- Parasitology Division, Children's Hospital "R Gutierrez" of Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Gonzalez NL, Moscatelli G, Moroni S, Ballering G, Jurado L, Falk N, Bochoeyer A, Goldsman A, Grippo M, Freilij H, Garcia Bournissen F, Chatelain E, Altcheh J. Long-term cardiology outcomes in children after early treatment for Chagas disease, an observational study. PLoS Negl Trop Dis. 2022 Dec 19;16(12):e0010968. doi: 10.1371/journal.pntd.0010968. eCollection 2022 Dec. PMID 36534647